CLINICAL TRIAL: NCT02630147
Title: Effects of Vanilla on Hypoxic Intermittent Events in Premature Infants
Acronym: Vanilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Paul Praud, MD, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1043
Record Dates: First submitted 2015-12-04; First posted 2015-12-15 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Premature Birth; Neonatal Hypoxic Conditions
Keywords: Late preterm; Vanilla; Hypoxic intermittent events
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vanilla, Then no vanilla night (Experimental): Participants were exposed to vanilla odor (2 mL of 2% vanillin on the bib, close to the face) on the first night (12-hour recording), and not exposed to vanilla on the third night (control night,12-hour recording)
  No intervention, no recordings were made on the second night
  Interventions: Other: Vanilla scent
- No vanilla, Then vanilla night (Experimental): Participants were exposed to the "control" condition on the first night, which consisted of no vanilla odor (12-hour recording), and then exposed to vanilla odor on the third night (2 mL of 2% vanillin on the bib, close to the face;12-hour recording)
  No intervention, no recordings were made on the second night
  Interventions: Other: Vanilla scent

INTERVENTIONS:
Other: Vanilla scent — A 12-hour continuous recording for monitoring hemoglobin oxygen saturation, electrocardiogram and respiratory movements will be performed while the infant is exposed to vanilla scent (from vanilla solution on the infant's pyjamas).

SUMMARY:
The purpose of this study is to evaluate the effect of vanilla odor on hypoxic intermittent events in premature infants born between 32.0 and 33.6 weeks of gestational age.

DETAILED DESCRIPTION:
A weekly screening will be done on all new hospitalized infants at the neonatal care unit of the CHUS born between 32.0 and 33.6 weeks of gestational age. At the beginning of their 2nd week in the neonatal care unit, infant's medical record will be consulted for inclusion and exclusion criteria. At this moment, no information will be noted. Then, team research will discuss with neonatologist to have their opinion concerning the inclusion of a patient in the study. If they agree, the doctor or the nurse having a therapeutic link with the infant will ask parents' infant if they agree to meet the research team to discuss about the research project. Once the agreement will be obtained, parents will be approached by a member of the research team. Project will be explained, questions will be answered and consent form will be obtained. When an infant will be enrolled in the study, a code will be attributed to him and a randomization will established the order of the intervention.

Option A) night 1: a 12h cardiorespiratory recording with vanilla, night 2: no recording and night 3: a 12h cardiorespiratory recording without vanilla OR Option B): night 1: a 12h cardiorespiratory recording without vanilla, night 2: no recording and night 3: a 12h cardiorespiratory recording recording with vanilla.

All data will be entered in a secured database and a double checked will be done by team members to assess the accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 30.0 and 34.0 weeks of gestational age;
* Postnatal age between 3 and 4 weeks;
* No current respiratory or ventilatory support;
* Stable state for at least the last 48 hours;
* Parental consent to enroll in the study.

Exclusion Criteria:

* Respiratory diseases other than apnea;
* Intraventricular hemorrhage grade 3 or 4 OR leukomalacia;
* Chromosomal abnormality;
* Congenital malformations which may result in cardiorespiratory or neurodevelopmental abnormality;
* Clinical deterioration during the study.

Ages: 3 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Praud, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Nicu - Chus, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All results will be made available with other researchers on demand, upon reasonable requests
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Available if requested, up to 2023
Access Criteria: Similar study protocol

REFERENCES:
- [Background] Brockmann PE, Poets A, Poets CF. Reference values for respiratory events in overnight polygraphy from infants aged 1 and 3months. Sleep Med. 2013 Dec;14(12):1323-7. doi: 10.1016/j.sleep.2013.07.016. Epub 2013 Oct 14. PMID 24211071
- [Background] Nunez J, Cristofalo E, McGinley B, Katz R, Glen DR, Gauda E. Temporal association of polysomnographic cardiorespiratory events with GER detected by MII-pH probe in the premature infant at term. J Pediatr Gastroenterol Nutr. 2011 May;52(5):523-31. doi: 10.1097/MPG.0b013e3181fa06d7. PMID 21502823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for eligibility and recruited in the neonatal care unit of the University of Sherbrooke Hospital Center, Canada, from November 2015 to February 2019.
Pre-assignment Details: Every baby was his own control (cross-over design)
  The aim was to get at least 30 enrolled newborns to have more than 20 valid recordings.
  We enrolled a total of 32 patients. 5 babies were withdrawed before recordings. This gave us 27 complete and analyzable recordings.
Groups:
- Vanilla, Then no Vanilla Night: Intervention = exposition to vanilla scent A quantity of 2 ml of a saturated vanilla solution (2% vanillin) will be applied on premature pyjamas infant's, close to his face (on each shoulder and on the upper chest).
  Vanilla scent: A 12-hour continuous recording for monitoring hemoglobin oxygen saturation, electrocardiogram and respiratory movements will be performed while the infant is exposed to vanilla scent (from vanilla solution on the infant's pyjamas).
  In addition, a 3-hour polysomnography will be done in a sub-sample on the morning following the night recording with vanilla solution.
- No Vanilla, Then Vanilla Night: The only difference with the experimental arm is the absence of vanilla (usual, standard care)
Period: First Intervention (First Night)
Arm/Group | Vanilla, Then no Vanilla Night | No Vanilla, Then Vanilla Night
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Washout, no Intervention (Second Night)
Arm/Group | Vanilla, Then no Vanilla Night | No Vanilla, Then Vanilla Night
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Second Intervention (Third Night)
Arm/Group | Vanilla, Then no Vanilla Night | No Vanilla, Then Vanilla Night
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vanilla, Then no Vanilla Night: First night: exposition to vanilla scent and recordings A quantity of 2 ml of a saturated vanilla solution (2% vanillin) were applied on premature pyjamas infant's, close to the face (on each shoulder and on the upper chest).
  Second night: No interventions, no recordings were made
  Third night: Control night, no vanilla, recordings for 12 hours
  Recordings: A 12-hour continuous recording for monitoring hemoglobin oxygen saturation, electrocardiogram and respiratory movements were performed.
- No Vanilla, Then Vanilla Night: First night: no exposition to vanilla scent, recordings (control night)
  Second night: No interventions, no recordings were made
  Third night: Vanilla exposition, with 2 ml of a saturated vanilla solution (2% vanillin) applied on premature pyjamas infant's, close to the face (on each shoulder and on the upper chest). Recordings for 12 hours
  Recordings: A 12-hour continuous recording for monitoring hemoglobin oxygen saturation, electrocardiogram and respiratory movements were performed.
- Total: Total of all reporting groups
Arm/Group | Vanilla, Then no Vanilla Night | No Vanilla, Then Vanilla Night | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 24.57 (4.48) | 23.93 (3.61) | 24.26 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 6 | 10 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 13 | 27
Gestational age [Median (Full Range); unit: Weeks] | 32 [30 to 33] | 32 [30 to 33] | 32 [30 to 33]
Chronological age [Median (Full Range); unit: Days] | 23 [19 to 32] | 25 [17 to 29] | 24 [17 to 32]
Caffeine [Count of Participants; unit: Participants] — Number of participants that were being treated with caffeine at the time of the study.
  Prolonged apneas of prematurity and periodic breathing have been treated primarily with caffeine which, overall, is accepted as a safe respiratory stimulant at standard dosage, though it may have unwanted side effects and is not always efficient.
  Participants | 13 | 10 | 23
Weight [Mean (Full Range); unit: kg] | 1.595 [1.08 to 2.22] | 1.75 [1.18 to 2.27] | 1.67 [1.08 to 2.27]

OUTCOME MEASURES:

1. Primary Outcome: Desaturation Index
Description: Number per hour of oxygen saturation < 90% for at least 5 seconds
Time Frame: 12 hour period of recording on the night 1 and 3 of each participants, in which they are exposed to vanilla or no vanilla odor
Population: The population in each group consists of the total participants number (27), since all children were exposed to the vanilla odor on one night, and all children were exposed to the control treatment on another night. In other words, all children were both in the vanilla night group, and the control night group.
Measure: Mean (Standard Deviation); unit: Number of events
Groups:
- Night-vanilla: Intervention = exposition to vanilla scent A quantity of 2 ml of a saturated vanilla solution (2% vanillin) will be applied on premature pyjamas infant's, close to his face (on each shoulder and on the upper chest).
  Vanilla scent: A 12-hour continuous recording for monitoring hemoglobin oxygen saturation, electrocardiogram and respiratory movements will be performed while the infant is exposed to vanilla scent (from vanilla solution on the infant's pyjamas).
- Night-no Vanilla: The only difference with the experimental arm is the absence of vanilla (usual, standard care)
Arm/Group | Night-vanilla | Night-no Vanilla
Number analyzed (Participants) | 27 | 27
Number of events | 51.7 (22.0) | 56.9 (25.7)

2. Secondary Outcome: Percentage of Time of Oxygen Saturation Under 90%
Description: Percentage time in overall duration of oxygen saturation under 90%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of overall time
Arm/Group | Night-vanilla | Night-no Vanilla
Number analyzed (Participants) | 27 | 27
% of overall time | 1.8 (1.23) | 2.2 (1.6)

3. Secondary Outcome: Percentage of Time of Periodic Breathing
Description: Percent of time of the recording spent in periodic breathing or in apnea.
  A periodic beathing epoch was defined as a series of 3 episodes or more of apneas lasting at least 3 seconds and separated by less than 20 seconds of normal breathing
  Apneas were defined as the absence of respiratory movements for at least 20 seconds or for at least 2 breathing cycles with a decrease of at least 3% in SpO2
Time Frame: as for outcome 1
Population: The number of usable recordings was 11 out of the 27, because the of technical recordings issues
Measure: Mean (Standard Deviation); unit: % of overall time
Arm/Group | Night-vanilla | Night-no Vanilla
Number analyzed (Participants) | 11 | 11
% of overall time | 12.2 (12.4) | 8.7 (10.2)

4. Secondary Outcome: Time in Apnea
Description: Percent of time of the recording spent in apnea
Time Frame: as for outcome 1
Population: The number of usable recordings was 11 out of the 27, because the of technical recordings issues
Measure: Mean (Standard Deviation); unit: % of overall time
Arm/Group | Night-vanilla | Night-no Vanilla
Number analyzed (Participants) | 11 | 11
% of overall time | 0.99 (0.4) | 1.02 (0.5)

5. Secondary Outcome: Mean SpO2
Description: Mean value of oxygen saturation (%)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of SpO2
Arm/Group | Night-vanilla | Night-no Vanilla
Number analyzed (Participants) | 27 | 27
% of SpO2 | 98 (1.2) | 97.5 (1.5)

ADVERSE EVENTS:
Time Frame: The period when adverse events was observed was during the 3 nights period.
Description: The participants were observed for any clinical changes that could happen during the trial, over the 3 days. A close collaboration with the neonatal team was performed to monitor any impacts.
Arm/Group | Night-vanilla | Night-no Vanilla
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT02630147/Prot_SAP_000.pdf